CLINICAL TRIAL: NCT00126191
Title: Phase II Study of Intensive Chemotherapy and Rituximab in Burkitt Lymphoma
Brief Title: Intensive Chemotherapy and Rituximab in the Treatment of Burkitt Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed due to slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ann S. LaCasce, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-336
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-04

CONDITIONS: Burkitt Lymphoma; Non-Hodgkins Lymphoma; Atypical Burkitt Lymphoma
Keywords: Burkitt Lymphoma; atypical Burkitt lymphoma; Non-Hodgkin's Lymphoma; rituximab
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Methotrexate; Leucovorin; Ifosfamide; Etoposide; Cytarabine; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Risk (Experimental): Low-risk patients receive 3 cycles of regimen A.
  Regimen A:
  Rituximab (375 mg/m^2) on Days 1 and 3. Cyclophosphamide (800 mg/m^2) on days 1 and 2. Vincristine (1.4 mg/m^2) on days 1 and 10. Doxorubicin (50 mg/m^2) on Day 1. Methotrexate (3000 mg/m^2) on Day 10. Intrathecal Cytarabine (50mg) will be given on Day 1 and intrathecal methotrexate (12mg) will be given on Days 1 and 10.
  Leucovorin on days 11 and 12.
  Rituximab is given on Days 1 and 3 in cycle 1, and on Day 1 of all other cycles.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Methotrexate; Drug: Leucovorin; Drug: Cytarabine
- High Risk (Experimental): High-risk patients receive 4 alternating cycles of regimens A and B (A-B-A-B).
  Regimen A (as described earlier).
  Regimen B:
  Rituximab (375mg/m^2) on Day 1. Ifosfamide (1500mg/m^2) on Days 1-5. Mesna (275 mg/m^2) on Days 1-5. Etoposide (60mg/mg^2) on Days 1-5. Cytarabine (2 gm/m^2) twice a day on Days 1 and 2. Intrathecal methotrexate (12mg) on Day 5, and intrathecal methotrexate (50mg) on Day 3 (also on Day 1 for patients with central nervous system involvement).
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Methotrexate; Drug: Leucovorin; Drug: Ifosfamide; Drug: Etoposide; Drug: Cytarabine; Drug: Mesna

INTERVENTIONS:
Drug: Rituximab — Low Risk: Intravenously on Day 3 of the first cycle (One cycle is 14 days) then day 1 for next 2 cycles (Regimen A) High Risk: Regimen A followed by a 5-day cycle where rituximan is given on day 1
  Other Names: Rituxan
Drug: Cyclophosphamide — Low Risk/High Risk: Intravenously on day 1 and day 2 of a 14-day cycle for 3 cycles (regimen A)
  Other Names: Cytoxan
Drug: Doxorubicin — Low Risk/High Risk: Given on day 1 of a 14-day cycle for 3 cycles (regimen A)
  Other Names: Adriamycin, Rubex
Drug: Vincristine — Low Risk/High Risk: Given intravenously on day 1 and day 10 of a 14-day cycle for 3 cycles (regimen A)
  Other Names: Oncovin, vincristine sulfate
Drug: Methotrexate — Low Risk: Given on day 10 of a 14-day cycle for 3 cycles (regimen A) High Risk: Regimen A followed by methotrexate on day 3 and day 5 of a 5-day cycle
  Other Names: Rheumatrex, Trexall
Drug: Leucovorin — Low Risk/High Risk: Given on days 11, 12 and 13 of a 14-day cycle for 3 cycles (regimen A)
  Other Names: Folinic acid
Drug: Ifosfamide — High Risk: After Regimen A, Ifosomide given on days 1-5 of a 5 day cycle
  Other Names: Ifex
  Arms: High Risk
Drug: Etoposide — High Risk: After Regimen A, etoposide given days 1-5 of a 5-day cycle
  Other Names: Vepesid
  Arms: High Risk
Drug: Cytarabine — Low Risk: Given on days 1, 3, 5 and 10 of a 14-day cycle for 3 cycles (regimen A) High Risk: After regimen A, cytarabine given on days 1 and 2 of a 5-day cycle
  Other Names: Cytosar, Tarabine PFS
Drug: Mesna — High Risk: After regimen A, mesna is given on days 1-5 of a 5-day cycle
  Other Names: Mesnex
  Arms: High Risk

SUMMARY:
The purpose of this study is to learn more about how well a chemotherapy regime including rituximab works in treating patients with Burkitt or atypical Burkitt lymphoma.

DETAILED DESCRIPTION:
* Patients will be placed into one of two groups, "low risk" and "high risk". "Low risk" disease is defined as one area of disease measuring less than 10cm and a normal blood test called LDH (lactate hydrogenase). Patients not fitting the "low risk" criteria are considered "high risk".
* If the patient has "low risk" disease their treatment cycle consist of three cycles of A.
* If the patient has "high risk" disease they will receive Cycle A followed by cycle B which will then repeat.
* Cycle A consists of the drugs: rituximab, cyclophosphamide, oncovin, doxorubicin and methotrexate (R-CODOX-M). The treatment cycle is approximately 14 days. A spinal tap is performed on day 1 and day 3 of the cycle and the patient will be hospitalized until between day 11 and day 13. After the patient's blood counts return to normal(usually around day 21),the next round of treatment will occur.
* Cycle B consists of the drugs: rituximab, ifosfamide, VP-16 and ara-c (IVAC). The treatment cycle is approximately 5 days. A spinal tap is performed on day 4 and once blood counts return to normal the patient will start cycle A again.
* After the patient has finished the treatments, they will be re-evaluated with CT scans and PET scans to determine whether or not they are in remission. Every three months for two years, blood tests and CT and PET scans will be performed. Follow up after that will be every 6 months for two years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented Burkitt or atypical Burkitt according to World Health Organization (WHO) criteria.
* Pathology must be reviewed at the Brigham and Women's Hospital (BWH).
* Measurable or evaluable disease: Disease reproducibly measurable in two perpendicular dimensions on exam, computed tomography (CT), radiograph, or magnetic resonance imaging (MRI). Disease present on bone marrow biopsy will be considered as evaluable disease.
* The following may not be used as the sole site of measurable or evaluable disease: *ascites, *pleural effusion, *bone lesion or *central nervous system (CNS) disease.
* Age > 18
* Laboratory data (within 2 weeks of study registration):

  * ANC > 1500/ul;
  * platelet > 100,000/ul;
  * creatinine < 1.5 X normal;
  * creatinine clearance > 60 ml/min;
  * bilirubin < 1.5 X normal;
  * AST and ALT < 2.5 X normal;
  * alkaline phosphates < 3 X normal;
  * HIV negative;
  * cardiac ejection fraction > 50%.

Exclusion Criteria:

* Previous chemotherapy or radiation therapy. Steroids of less than 72 hours duration for impending oncologic emergency are allowed.
* Uncontrolled bacterial, fungal, or viral infection.
* Concomitant malignancy excluding carcinoma in situ of the cervix and basal cell carcinoma of the skin.
* Serious comorbid disease. Clinically significant pulmonary symptomatology. In patients with a history of symptomatic pulmonary disease, pulmonary function tests (PFTs) should document an forced expiratory volume at 1 second (FeV1), forced vital capacity (FVC), and total lung capacity (TLC) of > 60% predicted and carbon monoxide diffusing capacity of the lung (DLCO) of > 50% predicted. No clinically significant cardiac symptomatology. The cardiac ejection fraction must be > 50%.
* Pregnancy. All males and females with reproductive potential must consent to use an effective form of contraception while on study.
* Major surgery within the previous 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann S. La Casce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This BL protocl was IRB approved 01/18/05, activated 7/18/05. Participants were identified either in the outpatient clinic at DFCI or while admitted to our partner inpatient hospital, Brigham & Women's Hospital. The study was closed to accrual 6/2/08 due to slow accrual.
Pre-assignment Details: Participants with previous chemotherapy or radiation, uncontrolled infection, concomitant malignancy (some exclusions), serious comorbid disease, pregnancy, and HIV+ were excluded. Subjects stratified according to risk: Single focus disease <10cm and normal LGH=low risk, all others high risk.
Groups:
- Low Risk: Regimen A. Single focus of disease less than 10 cm in greatest dimension and a normal LDH. Participants at low risk received three cycles of Regimen A (AAA).
- High Risk: Regimen A followed by Regimen B. Cycles A and B will then be repeated (ABAB).
Period: Overall Study
Arm/Group | Low Risk | High Risk
Started | 2 | 8
Completed | 2 | 6 (1 pt off study during cycle 1 due to toxicity)
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk | High Risk | Total
Number analyzed (Participants) | 2 | 8 | 10
Age, Categorical [Count of Participants; unit: Participants] — IRB approved deviation to register 1 patient at age 17.
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 1 | 8 | 9
    >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 1 | 8 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rates (CR and PR) in Adults With Burkitt/Atypical Burkitt
Description: Complete Response (CR): Disappearance of all measurable or evaluable disease confirmed.
  Partial Response (PR): Reduction of 50% or greater in the sum of the products of the perpendicular diameters of all measurable.
  Of 8 High Risk participants, 7 met the primary response outcome. 1 High Risk participant did not meet protocol defined primary outcome response and died two months following enrollment.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Low Risk | High Risk
Number analyzed (Participants) | 2 | 8
participants | 2 | 7

2. Secondary Outcome: Disease Free Survival
Description: Participants are followed after completion of protocol therapy until disease progression to determine disease free survival.
Time Frame: Until disease progression up to 120 months
Population: One low-risk participant was lost to follow-up after 48 months of disease free survival.
Measure: Mean (Full Range); unit: Months
Arm/Group | Low Risk | High Risk
Number analyzed (Participants) | 1 | 8
Months | 84 [84 to 84] | 52 [2 to 83]

ADVERSE EVENTS:
Description: Grade 4 hematologic toxicities were not considered to be serious adverse events in this Burkitts Lymphoma study. Hospitalization without accompanying SAE did not constitute SAE for this study.
Arm/Group | Low Risk | High Risk
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/8
Other Adverse Events (participants affected / at risk) | 0/2 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk (N=2) | High Risk (N=8)
Bilirubin (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hyperuricemia (Endocrine disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No